CLINICAL TRIAL: NCT03751618
Title: Prospective Study, Monocentric, Randomized, Double Blind Evaluating the Non Inferiority of Non Capsular Suture in Arthroscopic Treatment of Cam or Mixed-type Femoroacetabular Impingement Without Hip Dysplasia
Brief Title: Evaluation of Non Inferiority of Non Capsular Suture in Femoroacetabular Impingement Arthroscopic Treatment
Acronym: SUTURCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique de la Sauvegarde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2017-CSV-001
Record Dates: First submitted 2018-07-03; First posted 2018-11-23 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2018-11

CONDITIONS: Femoral Acetabular Impingement
Keywords: Hip arthroscopy; capsular suture; Femoral Acetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, randomized, double blind study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsular suture (Experimental): Capsular suture at the end of hip arthroscopy
  Interventions: Procedure: Hip arthroscopy
- No capsular suture (Active Comparator): No capsular suture at the end of hip arthroscopy
  Interventions: Procedure: Hip arthroscopy

INTERVENTIONS:
Procedure: Hip arthroscopy — Suture will be realized with two simple suture knots (non resorbable suture material). These suture knots will be performed at the end of hip arthroscopy. Correct capsular suture will be controlled under arthroscopy video.
  Patients randomized in control arm will not received capsular suture at the end of the procedure.

SUMMARY:
Since last past decade, arthroscopic hip surgery proved its efficacy in femoroacetabular impingement treatment. However, no consensus exist concerning capsular suture or not. According to capsular incision size, articular instability can persist if no suture is performed. In contrast, tightly suture can cause post-operative joint stiffness.

This study aims to evaluate the non inferiority of non capsular suture after hip arthroscopy treatment of cam or mixed-type femoroacetabular impingement, without hip dysplasia, after 2 years follow-up.

DETAILED DESCRIPTION:
Main Objective :

Non inferiority evaluation of non capsular suture after hip arthroscopy treatment of cam or mixed-type femoroacetabular impingement, without hip dysplasia, after 2 years follow-up.

The primary study endpoint is the patient reported outcomes (HAGOS score; iHOT-12 and MHHS) at 2 years follow-up.

Secundary objectives :

* Clinical results at 6 month and 1 year follow-up
* Specific complications occuring and frequences
* Patient quality of life,
* The return to sport,
* Sport level after surgery compare to sport level before surgery
* Pain

ELIGIBILITY:
Inclusion Criteria:

* patient < 18 years old
* Patient who can be followed for 2 years
* Patient with confirmed diagnostic of femoroacetabular impingement came or mixed-types, without dysplasia and with VCE angle > 25°, without prearthrosic lesion and Tonnis 0 ou Tonnis 1, radiographic assement
* Patient must sign an informed consent form indicating that he or she understands the purpose of procedure required for the study and accepts to participate in the study.
* Patient affiliated to a social security system

Exclusion Criteria:

* Patient with no wittren informed consent
* Patient presenting osteoarthritis (Tonnis stage 2) or only pincer impingement
* Hyperlaxity
* Dysplasia (VCE <25°)
* Patient already underwent hip arthroscopy
* Patient already underwent previous hip surgery
* Patient needing bilateral hip arthroscopy < 2 years
* Persons deprived of their freedom or under guardianship or incapable of giving consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
patient reported outcomes (questionnaires) | 2 years
  HAGOS score

SECONDARY OUTCOMES:
patient reported outcomes (questionnaires) | 6 months
  modified Harris Hip Score
patient reported outcomes (questionnaires) | 1 year
  iHOT-12

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France